CLINICAL TRIAL: NCT03025178
Title: External Validation of Predictive Formula for Optimal Insertion Depth of Left Internal Jugular Venous Catheter in Infants
Brief Title: Optimal Insertion Depth of Left Internal Jugular Vein Catheter in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H1701-038-821
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Central Venous Catheter; Infant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Central venous catheterization (Experimental): Central venous catheterization will be performed using 4Fr central venous catheter at left internal jugular vein in infant. The tip of central venous catheter will be confirmed by transthoracic echocardiography. The actual insertion depth of central venous catheter will be compared to the predicted insertion depth derived from two calculation methods using height and the distance between the anatomical landmarks.
  Interventions: Procedure: 4Fr central venous catheter insertion

INTERVENTIONS:
Procedure: 4Fr central venous catheter insertion — The central venous catheter is placed at left internal jugular vein in infant, and its tip is confirmed by transthoracic echocardiography.

SUMMARY:
We previously performed a study to create formula for the optimal insertion depth of left internal jugular vein catheter in infant, which was registered at cris.nih.go.kr. We found that two calculation methods using height and the distance between landmarks (0.11 × height (cm) + 0.19 and 1.02 × I-A-B (cm) + 1.55, where I was insertion point of needle, A was the most prominent point of the sternal head of the left clavicle, and B was the midpoint of the perpendicular line drawn between the sternal head of the right clavicle and an imaginary line between the nipples) were clinically feasible to determine the insertion depth of left internal jugular vein catheter. In this study, we will compare the actual insertion depth with the insertion depth determined from above two calculation methods in other 46 infants.

DETAILED DESCRIPTION:
determine the optimal insertion depth of left internal jugular vein catheter in infants

ELIGIBILITY:
Inclusion Criteria:

* An infant requiring a central venous catheter during surgery

Exclusion Criteria:

* Extracardiac vascular anomaly
* Dextrocardia
* Anatomical abnormality in neck and thorax

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
The actual insertion depth of central venous catheter | About 5 minutes during central venous catheterization (10 minutes after anesthetic induction)
  The actual insertion depth of central venous catheter placed at left internal jugular vein

SECONDARY OUTCOMES:
The differences between the actual insertion depth and the predicted insertion depth derived from two calculation methods | About 5 minutes during central venous catheterization (10 minutes after anesthetic induction)
  The differences between the actual insertion depth and the predicted insertion depth derived from two calculation methods

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided